CLINICAL TRIAL: NCT03482063
Title: The Effects of 12 Weeks Supplementation With a B-vitamin and Herbal Supplement on Neurocognitive Function and Mood: The Memory + Focus Clinical Trial (MAST - Memory and Attention Supplement Trial)
Brief Title: The Effects of 12 Weeks Supplementation With a B-vitamin and Herbal Supplement on Neurocognitive Function and Mood
Acronym: MAST
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Swisse Wellness Pty Ltd (Industry)
Collaborators: Swinburne University of Technology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: MAST
Record Dates: First submitted 2018-03-14; First posted 2018-03-29 (Actual); Last update posted 2020-03-18 (Actual); Status verified 2020-03

CONDITIONS: Neurocognitive Function; Mood
Keywords: B vitamin; herbal supplement; attention

STUDY DESIGN:
Intervention Model Description: Randomised, placebo-controlled, double-blind, parallel groups design
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Swisse Ultiboost Memory + Focus (Experimental): two tablets daily, one tablet during or immediately after breakfast, and one tablet during or immediately after lunch, for the duration of the trial period
  Interventions: Dietary Supplement: Swisse Ultiboost Memory + Focus
- Placebo (Placebo Comparator): two tablets daily, one tablet during or immediately after breakfast, and one tablet during or immediately after lunch, for the duration of the trial period
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Swisse Ultiboost Memory + Focus — B vitamins help energy release, help with metabolism of food into energy, assist energy production and vitality.
  Vitamin B5 helps support normal mental performance. Brahmi, Ginkgo, Vitamin B12 and B3 help support brain function. Ginkgo helps maintain healthy circulation and delivery of oxygenated blood to the brain.
  Brahmi supports memory function and recall. Vitamin B5, B6 are important for adrenal function, assist adrenal glands during stress periods.
  Vitamin B2, B3, B5, B6, B12 help relieve tiredness and fatigue.
  Arms: Swisse Ultiboost Memory + Focus
Other: Placebo — riboflavin (2.2mg)
  Arms: Placebo

SUMMARY:
The aim of the present study is to evaluate chronic supplementation with Swisse Ultiboost Memory + Focus over a 12 week period on memory in individuals with optimal and sub-optimal nutrient profiles.

DETAILED DESCRIPTION:
This study will have two co-primary outcomes; one each to measure memory and focus. Short term memory will be measured by the spatial working memory task from the Swinburne University Computerised Cognitive Assessment Battery. Focus will be measured by the incongruent version of the stroop colour-word task from the Swinburne University Computerised Cognitive Assessment Battery. Through investigations of blood vitamin markers, biomarkers of inflammation and neuroimaging techniques, this study aims to provide insight to the mechanisms through which the supplement is acting.

This study is a phase II clinical trial, which will follow a randomised, placebo-controlled, double-blind, parallel groups design. One hundred and forty participants will complete a 12 week intervention, which will involve three testing visits to Swinburne University, as well as in-home mood assessments. Of these, 60 participants will also complete an MRI component. Participants will be randomly allocated to one of two groups; one receiving active supplementation of Swisse Ultiboost Memory + Focus, and the other receiving a placebo formulation.

Prior to participants being enrolled in the study a telephone screening interview will be completed, to reduce the likelihood of ineligible participants attending study visits. Eligible participants will complete three study visits; a Screening and Practice visit (V0), Baseline Visit (V1), and the Final Visit (V2). The participant's baseline visit (V1) will be scheduled within two weeks of their screening and practice visit (V0). The participant's final visit (V2) will be scheduled 12 weeks (± 3 days) from the baseline visit (V1). Therefore, it is anticipated that participation in the trial will last a maximum of 14 weeks.

For the 12 week supplementation period between their baseline (V1) and final (V2) visits, participants will be instructed to consume one tablet, twice a day, of either Swisse Ultiboost Memory + Focus or placebo, with a meal. Participants will be requested to abstain from the treatment on the day of their final visit.

Participants will also be required to complete online mood assessments in their home, twice a week for the duration of the 12 week supplementation period. Two laboratory assessment points will be measured, at baseline (V1) and at the final visit (V2). Twenty four in-home assessment points will be measured, twice a week during participation in the study.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy males and females aged between 40 and 65 years
2. Non-smokers
3. English speaking
4. Not currently being treated for anxiety, depression or psychiatric disorders (if treatment was >2 years ago, can include)
5. Not suffering from cognitive impairment
6. No history of or currently suffering from neurological conditions (Epilepsy, Parkinsons, stroke, serious head trauma), cardiac diseases or diabetes requiring medication
7. Not taking any medication, herbal extracts, vitamin supplements or illicit drugs which might reasonably be expected to interfere with cognition or mood for 4 weeks prior to (and duration of) study, as defined by the exclusion list (Appendix 9)
8. No health conditions that would affect absorption of food, including the following: food allergies, impaired kidney function , liver disease (Hepatitis C, cirrhosis) and/or gastrointestinal diseases (e.g. Inflammatory bowel disease (Ulcerative Colitis, Crohn's Disease), coeliac disease, peptic ulcers)
9. Right handed (MRI component only)
10. Not hypertensive (systolic < 160 mm Hg and/or diastolic < 100 mm Hg at rest)
11. Not misusing substances
12. Have internet access in the home
13. Normal or corrected vision and normal colour vision
14. Not currently participating, or has not participated in another study investigating a nutraceutical supplement within the past 4 weeks
15. Not currently pregnant or lactating (for female participants of child bearing potential, the use of effective contraceptive method(s) for birth control for the duration of the study)
16. Willing and able to provide written informed consent.
17. Understands and is willing and able to comply with all study procedures.

Exclusion Criteria:

1. Chronic health condition
2. Smoker
3. Non-English speaking
4. Treatment for anxiety, depression (Becks Depression Inventory score ≥20 to be confirmed at screening visit) or other psychiatric conditions within the past 2 years
5. Suffering from cognitive impairment, dementia, Alzheimer's disease and/or a score of <24 on the Mini-Mental State Examination (to be confirmed at screening visit)
6. Neurological conditions (Epilepsy, Parkinsons, stroke, serious head trauma), cardiac diseases or diabetes requiring medication
7. Use of concomitant medications and/or vitamin supplements that could have cognitive or mood effects in the 4 weeks preceding the baseline visit, as defined by the exclusion list (Appendix 9)
8. Health conditions that would affect absorption of food, including the following: food allergies, impaired kidney function, liver disease (Hepatitis C, cirrhosis) and/or gastrointestinal diseases (e.g. Inflammatory bowel disease (Ulcerative Colitis, Crohn's Disease), coeliac disease, peptic ulcers)
9. Left handed (MRI participants only)
10. Blood pressure consistent with uncontrolled hypertension, (systolic > 160 mm Hg and/or diastolic > 100 mm Hg at rest)
11. Alcohol or substance abuse. Alcohol abuse is defined as >14 drinks per week.
12. Hypersensitivity to the investigational product or any of the active/inactive ingredients
13. Currently taking Warfarin
14. Currently participating, or has participated in another study investigating a nutraceutical supplement within the past 4 weeks
15. People with metal implants, pacemaker or aneurism clip (MRI participants only)
16. Currently pregnant or lactating
17. Any condition which may interfere with the subject's ability to perform assessments (e.g. claustrophobia for the MRI arm, dyslexia, colour blindness)

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 141 (Actual)
Dates: Start 2018-06-18 (Actual); Primary Completion 2020-01-09 (Actual); Study Completion 2020-01-09 (Actual)

PRIMARY OUTCOMES:
Changes in short term memory, as measured by the spatial working memory task from the Swinburne University Computerised Cognitive Assessment Battery. | 12 weeks
  In each trial participants are presented with a 4x4 white grid on a black background, with six grid positions containing white squares. Participants are given 3 seconds to remember where the white squares are located. The grid became blank and a series of four white squares were sequentially displayed in various grid positions for 2-seconds each. Participants responded with a yes/no response to indicate whether each square matched a position that was originally filled. In total, participants complete 14 trials, each of which are separated by a blank screen displayed for 2-seconds. Each trial was set such that two out of the four locations in the response series corresponded to the original grid locations, and two did not. The task requires participants to hold spatial information in working memory.
Changes in focus, as measured by the incongruent version of the stroop colour-word task from the Swinburne University Computerised Cognitive Assessment Battery | 12 weeks
  The test consists of congruent and incongruent trials blocks. Stimulus words are randomly presented (RED, BLUE, GREEN, YELLOW), printed in colours either congruent or incongruent with the written word. Participants are asked to respond by pressing one of four buttons corresponding to the colour of the print while ignoring the written word. The tasks are participant-paced, meaning that as soon as a participant responds to a word, they are presented with the next word. The incongruent trial will be used as a measure of selective attention as participants are required to selectively attend to the print colour of the written word, while inhibiting the automatic reading of the written word

SECONDARY OUTCOMES:
Simple reaction time component of the Swinburne University Computerised Cognitive Aging Battery (SUCCAB) | 12 weeks
  Participants respond with a right button press to the appearance of a single white square at the centre of the screen. Thirty targets are presented with a randomized inter-stimulus interval (ISI) to avoid anticipation effects.
Choice reaction time component of the Swinburne University Computerised Cognitive Battery (SUCCAB) | 12 weeks
  Participants respond with a left (blue) or right (red) button press to the appearance of a blue triangle or red square respectively. Presentation order and ISI are randomized to avoid anticipation effects.
Immediate/Delayed Recognition component of the Swinburne University Computerised Cognitive Battery (SUCCAB) | 12 weeks
  Participants are asked to study a series of 40 abstract images presented serially in the centre of the screen for 3-seconds each with no ISI. On completion, another series of images are presented, half of which were from the studied series and half that are new (Immediate condition). Participants indicate with a right (yes) or left (no) button press whether or not they recognized the image from the studied series. This task is repeated at the end of the testing session with the remaining 20 images from the studied series and another 20 new images (Delayed condition).
Stroop Colour-Word component of the Swinburne University Computerised Cognitive Battery (SUCCAB) | 12 weeks
  he test consists of two congruent and two incongruent trials, presented alternately. Stimulus words are randomly presented (RED, BLUE, GREEN, YELLOW) in either congruent or incongruent colours for 1.7-seconds, with an ISI of 0.5-seconds. Participants responded by pressing one of four buttons corresponding to the colour of the word, irrespective of what the word read. This task is used as a measure of executive function and more specifically inhibition; participants have to inhibit the automatic reading response.
Contextual memory component of the Swinburne University Computerised Cognitive Battery (SUCCAB) | 12 weeks
  A series of 20 everyday images are presented at the top/bottom/left/right of the screen for 3-seconds each with no ISI. On completion of the series the same images are displayed again in randomized order in the centre of the screen for 2-seconds each with no ISI. Participantsrespond with a top/bottom/left/right button press to indicate the original location of each image. The task requires participants to recall the spatial context of the original presentation and was used as a measure of episodic memory.
Serial Threes Subtraction component of the Cognitive Demand Battery | 12 weeks
  The participant is required to count backwards in threes from a random starting number between 800 and 999. The starting number is presented on the computer screen, and then is cleared by the first response. Participants are instructed to respond as quickly and as accurately as possible using computer keyboard keys. The participant completes the task over a period of two minutes.
Serial Sevens Subtraction component of the Cognitive Demand Battery | 12 weeks
  The participant is required to count backwards in sevens from a random starting number between 800 and 999. The starting number is presented on the computer screen, and then is cleared by the first response. Participants are instructed to respond as quickly and as accurately as possible using computer keyboard keys. The participant completes the task over a period of two minutes.
Rapid Visual Information Processing component of the Cognitive Demand Battery | 12 weeks
  A series of digits are presented in the centre of the screen at the rate of 100 per minute. The participant is required to detect three consecutive ascending odd or three consecutive ascending even digits. The participant responds to the detection of a target string by pressing the 'space bar'. The task is continuous for five minutes, with eight target strings presented each minute. This task is used as a measure of processing speed.
Perceived Stress Scale (PSS) | 12 weeks
  The PSS measures the extent to which respondents have perceived events in their life as stressful over the last month. There are 14 items, each scored on a 5-point scale ranging from 'never' to 'very often'. Seven of these items are positively stated items, and therefore they are reverse scored. Higher scores on the PSS are associated with higher levels of perceived stress.
Profile of Mood States (PROMS) | 12 weeks
  The POMS requires participants to indicate the degree to which they have identified with 65 mood-related adjectives over the past week. Each item is on a 5-point scale from 'not at all' to 'extremely'. Items are summed into six factors; Tensio n-Anxiety, Confusion-Bewilderment, Anger-Hostilit y, Depressio n-Dejection, Fatigue-Inertia and Vigor-Activit y.A Total Mood Disturbance (TMD) score is computed as the sum of the first 5 factors minus Vigor-Activity. High scores indicate greater mood disturbance on all scales except Vigor-Activity.
The Depression, Anxiety and Stress Scale (DASS) | 12 weeks
  The DASS measures comprises of 21 items that pertain to affect- related symptoms for three sub-factors: depression, anxiety and stress. Participants must respond to each item to reflect their experiences over the past week. Each item is on a 4-point scale fro m 0 to 3, with a total range of scores from 0 to 63. Higher scores indicate a higher degree of dysfunction and less desirable affect experience. A score of zero does not indicate positive mood, but rather the lack of presence of negative mood state symptoms. The DASS is considered relevant for both clinical and non-clinical populations as some experience of such symptoms is considered normal in day to day life.
State-Trait Anxiety Inventory - State Subscale (STAI-S) | 12 weeks
  The State-Trait Anxiety Inventory (STAI) contains two subscales; one that measures the transient experiences of anxiety (STAI-S) and the other measures the more stable personality characteristic (STAI-T). The state subscale (STAI-S) contains 20 items, asking participants about to respond with how they are feeling 'right now', ranging from 'not at all' to 'very much so'. The total range of scores is from 20 to 80, with higher scores indicating higher levels of anxiety.
Bond-Lader Visual Analogue Scales (VAS) | 12 weeks
  This task comprises of 16 100mm lines anchored at either end by antonyms. Participants must mark their current subjective state between the antonyms on each line, bearing in mind that each end of the scale represents an extreme. Each line is scored as millimetres to the mark from the negative antonym. From the scores, a factor analysis can isolate three factors; 'alertness', 'calmness' and 'contentedness'. Scores for each factor represent the unweighted average number of millimetres from the negative antonym for the individual scales contributing to the factor.
Stress, Anxiety, Mental Fatigue, Concentration and Mental Stamina Visual Analogue Mood Scales (VAMS) | 12 weeks
  The following scales will ask the participant to rate their subjective experiences of stress, fatigue, concentration and stamina in the present moment. In each case, participants will rate their subjective feeling on a 100mm visual analogue scale, and be required to mark the line as a response to reflect their current subjective state: Stress, anxiety, mental fatigue, concentration, mental stamina.
Prospective and Retrospective Memory Questionnaire (PRMQ) | 12 weeks
  The PRMQ is a self-rated measure of prospective and retrospective memory slips in everyday life. It consists of sixteen statements, half which relate to prospective memory failures, and the other half relate to retrospective failures. The participant must respond with how often each statement applies to them. Items are scored in a likert format with response options from 'very often' to 'never'.
Chalder Fatigue Scale (CFS) | 12 weeks
  The CFS is a self-rated measure of fatigue severity over the past week. The scale consists of 14 items, eight relating to physical symptoms and six questions relating to mental fat igue. Items are scored in a likert format with response options ranging from 'better than usual' to 'much worse than usual'.
Subjective Experience Survey | 12 weeks
  At the end of the study, participants will be asked the following qualitative questions: 1.While taking part in this study, have you experienced any positive changes in your physical or mental health (mood, stress, brain function) that you don't know the cause of or you think may be caused by the study tablets? 2.While taking part in this study, have you experienced any negative changes in your physical or mental health (mood, stress, brain function) that you don't know the cause of or you think may be caused by the study tablets? 3.While taking part in this study have you experienced any unusual changes (not necessarily good or bad) in your physical or mental health (mood, stress, brain function) that you don't know the cause of or you think may be caused by the study tablets? These questions are designed to capture any additional changes to cognition or mood that may not be picked up using the other questionnaires.
Biomedical measures | 12 weeks
  Participants will have fasting blood samples taken at the participant's baseline (V1) visit and their final (V2) visit. Blood samples will be collected by a qualified venepuncture technician or research nurse at the Centre for Human Psychopharmacology and securely stored in a freezer. All blood samples (with the exception of blood for essential fatty acid panel analysis) will sent to an Australian Clinical Labs pathology lab in Melbourne to be analysed. Samples used for essential fatty acid panel analysis will be sent to the University of Adelaide pathology lab to be analysed.
  Samples will be tested for: Vitamin B1, B2, B6, B12, Red Cell Folate and Homocysteine, high-sensitivity C-reactive protein, electrolytes, renal function, liver function and cholesterol.
  A medical investigator will assess the clinical significance of any abnormal values.
Neuroimaging | 12 weeks
  Participants who are consented for additional neuroimaging will undergo the following: functional magnetic resonance imaging, arterial spin labelling and diffusion tensor imaging.

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Pipingas, Principal Investigator — Swinburne University
Locations (1):
- Swinburne University of Technology, Hawthorn, Victoria, Australia

IPD SHARING:
Plan to Share IPD: No